CLINICAL TRIAL: NCT01363466
Title: Randomized Phase III Trial Evaluating the Impact of Hysterectomy After Chemoradiation Therapy for Stage IB2/II Cervical Cancer
Brief Title: Evaluation of Hysterectomy After Chemoradiation Therapy for Stage IB2/II Cervical Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: low recruitment
Sponsor: UNICANCER (Other)
Responsible Party: Professor Philippe MORICE, Institut Gustave Roussy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GYNECO 02/0108
Record Dates: First submitted 2011-05-05; First posted 2011-06-01 (Estimated); Last update posted 2011-06-01 (Estimated); Status verified 2011-05

CONDITIONS: Stage IB2 Cervical Cancer; Stage II Cervical Cancer; Adenocarcinoma; Squamous Cell Carcinoma; Adenosquamous Carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms; Adenocarcinoma; Carcinoma, Squamous Cell; Carcinoma, Adenosquamous | interventions — Hysterectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- with hysterectomy (Experimental)
  Interventions: Procedure: hysterectomy
- without hysterectomy (No Intervention)

INTERVENTIONS:
Procedure: hysterectomy
  Arms: with hysterectomy

SUMMARY:
GYNECO 02 hypothesis is that hysterectomy reduces the possibility of local or loco-regional relapse, especially in patient with a reduced metastatic risk and who received a local chemoradiation therapy with an increase of radiotherapy doses (45 grays).

ELIGIBILITY:
Inclusion Criteria:

* operable Stage IB2/II Cervical Cancer
* adenocarcinoma, squamous cell or adenosquamous carcinoma
* Patient between 18 and 70 years old
* No lombo-aortic lymph node invasion at baseline
* Previous 45 grays external pelvic radiation with concomitant chemotherapy (cisplatin 40 mg/m2/week corresponding to 5 cycles)
* Followed by a 15 grays utero-vaginal brachytherapy, eventually combined with a 6th cycle of chemotherapy (cisplatin 40 mg/m2)
* with a pelvic boost if lymph node or parametrial invasion
* No macroscopic residual tumor after 6 to 8 weeks after brachytherapy.

Exclusion Criteria:

* Other tumor histology (neuro-endocrine)
* Stage > II (FIGO 1995) at baseline
* Patient with remaining cervical cancer (after sub-total hysterectomy)

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2003-05; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Relapse free survival | from randomization to relapse or last contact (up to 3 years)
  There is a follow-up period of 3 years.

SECONDARY OUTCOMES:
Overall Survival | From randomisation to death or last contact (up to 3 years)
  There is a follow-up period of 3 years.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe MORICE, Pr, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (35):
- France (35):
  - Clinique Axium, Aix-en-Provence
  - Polyclinique du Parc Rambot, Aix-en-Provence
  - Clinique Sainte Thérèse de l'enfant Jésus, Amiens
  - Centre Hospitalier Universitaire, Amiens
  - Centre Paul Papin, Angers
  - Centre Hospitalier de Beauvais, Beauvais
  - Institut Bergonié, Bordeaux
  - Centre Hospitalier Nord Deux-Sèvres, Bressuire
  - Centre Hospitalier Universitaire de Brest, Brest
  - Centre Hospitalier Intercommunal, Créteil
  - Centre Georges-François Leclerc, Dijon
  - Centre Hospitalier de Fontainebleau, Fontainebleau
  - Hôpital Hotel-Dieu, Lyon
  - Centre Hospitalier Edouard Herriot, Lyon
  - Centre Hospitalier Lyon Sud, Lyon
  - Institut paoli Calmettes, Marseille
  - Centre Hospitalier Régional Universitaire La Timone, Marseille
  - Hôpital de la conception, Marseille
  - Centre Hospitalier Régional Universitaire Hôpital Nord, Marseille
  - Centre Hospitalier Universitaire - Hôpital Arnaud de Villeneuve, Montpellier
  - Centre Val d'Aurelle-Paul Lamarque, Montpellier
  - Centre hospitalier des Pays de Morlaix, Morlaix
  - Centre René Gauducheau, Nantes
  - Hôpital de la Source, Orléans
  - Hôpital des Diaconnesses, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Centre Hospitalier Universitaire Jean Bernard, Poitiers
  - Polyclinique de Courlancy, Reims
  - Clinique Mutualiste de la Sagesse, Rennes
  - Centre Universitaire Hospitalier- Hôpital Sud, Rennes
  - Centre Henri Becquerel, Rouen
  - Centre René Huguenin, Saint-Cloud
  - Institut Claudius Régaud, Toulouse
  - Centre Hospitalier Bretonneau, Tours
  - Institut Gustave Roussy, Villejuif